CLINICAL TRIAL: NCT03183596
Title: Optimal Injection Site for Serratus Anterior Plane Block in Reconstructive Breast Surgery (Randomized, Pilot Study)
Brief Title: Optimal Injection Site for Serratus Anterior Plane Block in Reconstructive Breast Surgery
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Principal investigator determination
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Christopher Godlewski, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: F000000000
Record Dates: First submitted 2017-06-07; First posted 2017-06-12 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Pain, Postoperative
Keywords: Deep Serratus Block; Reconstructive Breast Surgery; Superficial Serratus block
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Intervention Model Description: There has been no large, randomized study to define optimal location of injection based on analgesia and duration. Patients will be randomized to receive a "deep" Serratus Anterior Block (DSAB) where local anesthetic is deposited deep to the serratus or a "superficial" Serratus Anterior Block (SSAB) where the local anesthetic is placed between serratus and latissimus dorsi.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Deep Serratus Anterior Block (Active Comparator): Patients in the "deep" Serratus Anterior Block (DSAB) group will have 20-60cc of 0.25% bupivacaine and 2-4mg of dexamethasone deposited deep to the serratus. The investigator will then evaluate the difference based on pain scores, opiate consumption, length of hospital stay, as well as nausea and vomiting.
  Interventions: Drug: Bupivacaine; Drug: Dexamethasone
- Superficial Serratus Anterior Block (Active Comparator): Patients in the "superficial" Serratus Anterior Block (SSAB) group will have 20-60cc of 0.25% bupivacaine and 2-4mg of dexamethasone placed between serratus and latissimus dorsi. The investigator will then evaluate the difference based on pain scores, opiate consumption, length of hospital stay, as well as nausea and vomiting.
  Interventions: Drug: Bupivacaine; Drug: Dexamethasone

INTERVENTIONS:
Drug: Bupivacaine — 20-60cc of 0.25% Bupivacaine
  Other Names: Marcaine, Sensorcaine
Drug: Dexamethasone — 2-4mg of Dexamethasone
  Other Names: Ozurdex, Decadron, DexPak, Maxidex, Baycadron

SUMMARY:
The novel introduction of various chest wall blocks such as the Pecs I and II/modified Pecs blocks as well as the Serratus Anterior Plane Block have extended the application of perioperative regional anesthesia to provide analgesia for breast surgery. However, to our knowledge, there are no large studies that truly delineate the optimal injection site for the Serratus Anterior Plane Block.

DETAILED DESCRIPTION:
Analgesia for reconstructive breast surgery can be a challenging undertaking; these women have often been through painful mastectomy procedures coupled with the mental and physical discomfort of chemotherapy and its attendant side effects. Additionally, the surgery itself can provoke significant pain; often requiring extensive dissection of soft tissue and muscle to provide flap coverage as well the real discomfort of tissue expansion. The literature has described 2 possible injection sites for the Serratus Anterior Block, however, no study has defined optimal location based on analgesia and duration. Patients will be randomized to receive a "deep" Serratus Anterior Block (DSAB) where local anesthetic is deposited deep to the serratus or a "superficial" Serratus Anterior Block (SSAB) where the local anesthetic is placed between serratus and latissimus dorsi. The investigator will then evaluate the difference based on pain scores, opiate consumption, length of hospital stay, as well as nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing reconstructive breast surgery

Exclusion Criteria:

* Patients with allergies to the local anesthetic
* Patients who do no consent to regional anesthesia
* Patients in which serratus block would be contraindicated
* Patients whose anatomy preclude placement of the block

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Total Pain Score | baseline to 48 hrs postoperatively
  Collection of pain scores (VAS) until approximately 48 hours post-operatively

SECONDARY OUTCOMES:
Average Opioid consumption | 48 hrs postoperatively
  Average opioid consumption 48hrs postoperatively between study group and control
Length of Stay | baseline to 72 hrs post-operatively
  Number of days in the hospital
PONV Medications | baseline to 48 hrs post-operatively
  Mean time onset use of rescue PONV medications postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Godlewski, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Department of Anesthesiology and Perioperative Medicine, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No